CLINICAL TRIAL: NCT03534284
Title: Short and Long-Term Effectiveness of Existing Insomnia Therapies for Patients Undergoing Hemodialysis (Sleep-HD)
Brief Title: Short and Long-Term Effectiveness of Existing Insomnia Therapies for Patients Undergoing Hemodialysis
Acronym: Sleep-HD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rajnish Mehrotra, Section Head Nephrology, School of Medicine: Department of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004678; R01DK115468 (NIH)
Record Dates: First submitted 2018-05-01; First posted 2018-05-23 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Insomnia; End Stage Renal Disease
Keywords: Hemodialysis; Kidney disease; Trazodone; Cognitive behavioral therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Kidney Failure, Chronic; Kidney Diseases | interventions — Cognitive Behavioral Therapy; Trazodone

STUDY DESIGN:
Intervention Model Description: SLEEP-HD is a parallel group randomized controlled trial wherein 125 HD patients with chronic insomnia, treated in community-based dialysis facilities in Seattle and Albuquerque, will be randomized 1:1:1 over 31 months to 6-week treatment with telehealth CBT-I, trazodone, or medication placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigator, the participant, and the care provider will be blinded to the drug assignment (trazodone vs. placebo) for those subjects randomized into the medication intervention arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CBT-I (Active Comparator): Cognitive Behavioral Therapy for Insomnia sessions: a 30-minute treatment session once weekly for six weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Medication- Trazodone (Active Comparator): Trazodone (50-100 mg):
  Interventions: Drug: Trazodone
- Medication- Placebo (Placebo Comparator): Placebo (for trazodone)
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Once weekly treatment sessions for 6 weeks. The content of each of these sessions will be adapted to include changes in behavior during HD treatments (such as napping) and to help patients better adjust to treatment schedules. The CBT-I sessions will be delivered by a therapist face-to-face with the patient via a fully interactive video telehealth platform.
  Other Names: CBT-I
  Arms: CBT-I
Drug: Trazodone — trazodone tablet
  Other Names: Desyrel
  Arms: Medication- Trazodone
Drug: Placebo — Inactive pill manufactured to mimic trazodone tablets.
  Other Names: Placebo (for trazodone)
  Arms: Medication- Placebo

SUMMARY:
Insomnia is a common and distressing symptom for patients on hemodialysis (HD), and there is evidence for a much larger impact on the health of patients. Chronic insomnia is disrupted sleep that occurs at least three nights per week and lasts at least three months.

The SLEEP-HD study is a randomized open-label clinical trial to compare two types of treatment for insomnia in participants who have end-stage renal disease on HD, and who have been diagnosed with chronic insomnia. The two types of treatment involved in the study are Cognitive Behavioral Therapy for Insomnia (CBT-I) or treatment with a drug (trazodone vs placebo).

126 participants will be enrolled who are undergoing HD in two study locations (Seattle, Washington and Albuquerque, New Mexico).

DETAILED DESCRIPTION:
Most HD patients have significant impairments in quality of life, largely from the high frequency of disabling symptoms. Insomnia is one of the most frequently reported symptoms and studies of HD patients and/or other populations suggest that it is a significant contributor to other common symptoms and poor health outcomes. There are unique contributors to chronic insomnia in HD patients and these include the biologic effects of residual uremia after partial correction as is achieved with current dialysis technology, maladaptation to treatment schedules, and patients' napping during treatments.

There is a compelling need to identify effective treatments for insomnia in HD patients and the interventions being studied in this clinical trial, telehealth cognitive behavioral therapy for insomnia (CBT-I) and trazodone, have a strong scientific premise. If telehealth (web-based) CBT-I is effective for insomnia in HD patients, it will make a treatment that is presently inaccessible available to patients. Trazodone is widely used but the data on efficacy for insomnia are limited; no such data exist for HD patients.

SLEEP-HD is a parallel group randomized controlled trial wherein 125 HD patients with chronic insomnia, treated in community-based dialysis facilities in Seattle and Albuquerque, will be randomized 1:1:1 over 31 months to 6-week treatment with telehealth CBT-I, trazodone, or medication placebo.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing thrice-weekly maintenance hemodialysis for ≥ 3 months
* Able to speak English
* ISI score ≥ 10 at pre-screening with sleep disturbances for ≥ 3 nights per week for ≥ 3 months

Exclusion Criteria:

* Severe cognitive impairment on Mini-COG cognitive test (score < 3)
* Severe depression assessed by Patient Health Questionnaire (PHQ)-2 and if appropriate, PHQ-9
* Suicidal Ideation
* Alcohol abuse on CAGE alcohol assessment questionnaire (score ≥ 2) or substance abuse on Drug Abuse Screening Test (DAST)-10 questionnaire (score > 5)
* Severe restless leg syndrome
* Treatment with trazodone in the past one month
* Known allergy to trazodone (self-report or by chart review)
* Current treatment with monoamine oxidase inhibitors or in the preceding 14 days
* Current treatment with linezolid (self-report or by chart review)
* Current treatment with other drugs that are inhibitors of CYP3A4 (e.g., itraconazole, clarithromycin, voriconazole), or known to prolong QT interval including Class 1A antiarrhythmics (e.g., quinidine, procainamide) or Class 3 antiarrhythmics (e.g., amiodarone, sotalol), antipsychotic medications (ziprasidone, chlorpromazine, thioridazine), and quinolone antibiotics
* Pregnancy, or lactation, or women of childbearing potential not willing to use adequate birth control
* Life Expectancy < 3 months
* Expected to receive a kidney transplant or transition to home dialysis (peritoneal dialysis or home hemodialysis) within 6 months
* Any other condition that, in the opinion of the investigator, should preclude patient participation in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj Mehrotra, MD, Principal Investigator — University of Washington
Locations (1):
- Northwest Kidney Centers, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehrotra R, Cukor D, McCurry SM, Rue T, Roumelioti ME, Heagerty PJ, Unruh M. Effectiveness of Existing Insomnia Therapies for Patients Undergoing Hemodialysis : A Randomized Clinical Trial. Ann Intern Med. 2024 Feb;177(2):177-188. doi: 10.7326/M23-1794. Epub 2024 Jan 16. PMID 38224591
- [Derived] Unruh M, Cukor D, Rue T, Abad K, Roumelioti ME, McCurry SM, Heagerty P, Mehrotra R. Sleep-HD trial: short and long-term effectiveness of existing insomnia therapies for patients undergoing hemodialysis. BMC Nephrol. 2020 Oct 20;21(1):443. doi: 10.1186/s12882-020-02107-x. PMID 33081705

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 923 patients screened with Insomnia Severity Index (ISI). Of 411 identified as having insomnia (ISI score >=10),179 declined study participation and 106 met exclusion criteria.
Pre-assignment Details: 126 participants completed baseline measures before group assignment, including patient reported outcomes collected via Computer Assisted Telephone Interview (CATI) and nights using sleep aid on sedatives&hypnotics CRF. Most (115) also completed baseline Actigraphy, although this was not required for study entry (randomization).
Period: Overall Study
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Started | 43 | 42 | 41
Week 7 Primary Outcome | 39 | 41 | 40
Completed (Week 25 primary outcome) | 36 | 39 | 38
Not Completed | 7 | 3 | 3
Not completed — Death | 2 | 3 | 3
Not completed — Withdrawal by Subject | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo | Total
Number analyzed (Participants) | 43 | 42 | 41 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (15.2) | 56.2 (13.4) | 57.2 (12.7) | 58.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 19 | 63
  Male | 21 | 20 | 22 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 8 | 26
  Not Hispanic or Latino | 34 | 33 | 33 | 100
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 3 | 7
  Asian | 2 | 2 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2 | 4
  Black or African American | 9 | 9 | 9 | 27
  White | 28 | 27 | 23 | 78
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Time since starting dialysis, months [Median (Inter-Quartile Range); unit: months] | 26.4 [15.8 to 45.7] | 36.3 [19.6 to 58.2] | 28.2 [14.0 to 52.5] | 30.9 [15.5 to 52.4]

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI) Short-term
Description: summary score obtained from the ISI, measuring insomnia, range from 0 to 28. Higher score indicates greater insomnia, at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: The model used to estimate means at week 7 and week 25 included all time points (weeks 0, 4, 7, 13, 25). All N=126 participants had the outcome on at least one time point. Thus the model included all participants, even those missing outcome at week 7 or week 25.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 12.47 [10.68 to 14.26] | 11.97 [10.23 to 13.72] | 13.05 [11.29 to 14.82]
Statistical Analysis 1: Comparison: CBT-I vs Medication- Trazodone vs Medication- Placebo; Null hypothesis: average CBT-I=Trazodone=Placebo at week 7; Test type: Superiority; p = 0.6761, Mixed Models Analysis — 0.05 threshold for significance; no adjustment for multiple comparisons

2. Primary Outcome: Insomnia Severity Index (ISI) Long-term
Description: summary score obtained from the ISI, measuring insomnia, range from 0 to 28. Higher score indicates greater insomnia, at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 11.34 [9.28 to 13.41] | 12.2 [10.2 to 14.19] | 11.85 [9.83 to 13.88]
Statistical Analysis 1: Comparison: CBT-I vs Medication- Trazodone vs Medication- Placebo; Null hypothesis: average CBT-I=Trazodone=Placebo at week 25; Test type: Superiority; p = 0.8375, Mixed Models Analysis

3. Secondary Outcome: Patient-reported Outcomes (PRO) - Pittsburgh Sleep Quality Index - Short-term
Description: Score from Pittsburgh Sleep Quality Index, measuring sleep quality, range 0 to 21. Higher scores indicates worse sleep quality: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 9.44 [8.32 to 10.55] | 11.09 [10 to 12.18] | 12.39 [11.28 to 13.49]

4. Secondary Outcome: Patient-reported Outcomes (PRO) - Pittsburgh Sleep Quality Index - Long-term
Description: Score from Pittsburgh Sleep Quality Index, measuring sleep quality, range 0 to 21. Higher scores indicates worse sleep quality: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 9.15 [7.89 to 10.4] | 10.49 [9.26 to 11.71] | 9.95 [8.71 to 11.19]

5. Secondary Outcome: Patient-reported Outcomes (PRO) - Epworth Sleepiness Scale - Short-term
Description: Score from Epworth Sleepiness Scale, measuring sleepiness, range 0 to 24. Higher scores indicates greater sleepiness: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 7.67 [6.37 to 8.97] | 8.46 [7.19 to 9.74] | 7.5 [6.21 to 8.79]

6. Secondary Outcome: Patient-reported Outcomes (PRO) - Epworth Sleepiness Scale - Long-term
Description: Score from Epworth Sleepiness Scale, measuring sleepiness, range 0 to 24. Higher scores indicates greater sleepiness: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 7.27 [5.88 to 8.65] | 8.12 [6.76 to 9.47] | 7.94 [6.57 to 9.31]

7. Secondary Outcome: Patient-reported Outcomes (PRO) - FACIT Fatigue Scale- Short-term
Description: Score from FACIT Fatigue Scale, measuring fatigue, range 0 to 52. Higher scores indicates greater fatigue: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 32.55 [29.51 to 35.59] | 28.76 [25.77 to 31.75] | 28.5 [25.48 to 31.51]

8. Secondary Outcome: Patient-reported Outcomes (PRO) - FACIT Fatigue Scale- Long-term
Description: Score from FACIT Fatigue Scale, measuring fatigue, range 0 to 52. Higher scores indicates greater fatigue: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 32.65 [29.44 to 35.86] | 28.53 [25.39 to 31.68] | 30.7 [27.52 to 33.87]

9. Secondary Outcome: Patient-reported Outcomes (PRO) - Graded Chronic Pain Scale - Short-term
Description: Score from first item Graded Chronic Pain scale, measuring pain, range 0 to 10. Higher scores indicates greater pain: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
units on a scale | 4.50 [3.74 to 5.27] | 4.53 [3.78 to 5.29] | 4.21 [3.44 to 4.98]

10. Secondary Outcome: Patient-reported Outcomes (PRO) - Graded Chronic Pain Scale - Long-term
Description: Score from first item Graded Chronic Pain scale, measuring pain, range 0 to 10. Higher scores indicates greater pain: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
units on a scale | 4.14 [3.34 to 4.95] | 4.32 [3.53 to 5.11] | 4.80 [4.00 to 5.60]

11. Secondary Outcome: Patient-reported Outcomes (PRO) - Graded Chronic Pain Scale - Interference - Short-term
Description: Score from Second Item Graded Chronic Pain scale, measuring pain interference, range 0 to 10. Higher scores indicates greater interference from pain: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
units on a scale | 4.18 [3.32 to 5.05] | 4.07 [3.22 to 4.91] | 3.61 [2.75 to 4.46]

12. Secondary Outcome: Patient-reported Outcomes (PRO) - Graded Chronic Pain Scale - Interference - Long-term
Description: Score from Second Item Graded Chronic Pain scale, measuring pain interference, range 0 to 10. Higher scores indicates greater interference from pain: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
units on a scale | 3.88 [3.07 to 4.68] | 3.71 [2.93 to 4.50] | 4.30 [3.50 to 5.09]

13. Secondary Outcome: Patient-reported Outcomes (PRO) - Patient Health Questionnaire 9 - Short-term
Description: Score from Patient Health Questionnaire 9, measuring depression, range 0 to 27. Higher scores indicates greater depression: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 6.98 [5.47 to 8.49] | 7.93 [6.45 to 9.40] | 8.27 [6.78 to 9.75]

14. Secondary Outcome: Patient-reported Outcomes (PRO) - Patient Health Questionnaire 9 - Long-term
Description: Score from Patient Health Questionnaire 9, measuring depression, range 0 to 27. Higher scores indicates greater depression: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 6.61 [5.09 to 8.14] | 8.04 [6.55 to 9.53] | 7.34 [5.83 to 8.84]

15. Secondary Outcome: Patient-reported Outcomes (PRO) - Generalized Anxiety Disorder 7 Scale - Short-term
Description: Score from Generalized Anxiety Disorder 7 Scale, measuring anxiety, range 0 to 21. Higher scores indicates greater anxiety: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 5.18 [3.54 to 6.82] | 6.18 [4.58 to 7.79] | 7.04 [5.42 to 8.66]

16. Secondary Outcome: Patient-reported Outcomes (PRO) - Generalized Anxiety Disorder 7 Scale - Long-term
Description: Score from Generalized Anxiety Disorder 7 Scale, measuring anxiety, range 0 to 21. Higher scores indicates greater anxiety: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 5.27 [3.56 to 6.98] | 6.35 [4.67 to 8.02] | 6.29 [4.60 to 7.99]

17. Secondary Outcome: Patient-reported Outcomes (PRO) - Quality of Life Short Form 12 Scale - Physical Component Score - Short-term
Description: Score from Quality of Life Short Form 12 scale - Physical Component Score, measuring quality of life, range 0 to 100. Higher scores indicates better quality of life: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 31.87 [29.13 to 34.61] | 32.37 [29.66 to 35.08] | 32.80 [30.06 to 35.53]

18. Secondary Outcome: Patient-reported Outcomes (PRO) - Quality of Life Short Form 12 Scale - Physical Component Score - Long-term
Description: Score from Quality of Life Short Form 12 scale - Physical Component Score, measuring quality of life, range 0 to 100. Higher scores indicates better quality of life: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 33.21 [30.36 to 36.07] | 32.07 [29.28 to 34.85] | 31.85 [29.04 to 34.67]

19. Secondary Outcome: Patient-reported Outcomes (PRO) - Quality of Life Short Form 12 Scale - Mental Component Score - Short-term
Description: Score from Quality of Life Short Form 12 scale - Mental Component Score, measuring quality of life, range 0 to 100. Higher scores indicates better quality of life: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 49.53 [46.62 to 52.44] | 47.77 [44.90 to 50.65] | 48.29 [45.38 to 51.19]

20. Secondary Outcome: Patient-reported Outcomes (PRO) - Quality of Life Short Form 12 Scale - Mental Component Score - Long-term
Description: Score from Quality of Life Short Form 12 scale - Mental Component Score, measuring quality of life, range 0 to 100. Higher scores indicates better quality of life: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 50.44 [47.59 to 53.29] | 49.23 [46.45 to 52.01] | 51.38 [48.56 to 54.19]

21. Secondary Outcome: Cumulative Weekly Use of Sedatives/Hypnotics - Short-term
Description: This will be defined, as the number of days that the patient took a drug to help sleep, range from 0 to 7: at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
days | 1.65 [0.93 to 2.37] | 1.29 [0.66 to 1.92] | 1.01 [0.35 to 1.67]

22. Secondary Outcome: Cumulative Weekly Use of Sedatives/Hypnotics - Long-term
Description: This will be defined, as the number of days that the patient took a drug to help sleep, range from 0 to 7: at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 43 | 42 | 41
days | 1.58 [0.93 to 2.24] | 2.62 [1.69 to 3.56] | 2.42 [1.51 to 3.32]

23. Secondary Outcome: Objective Measure of Sleep - Short-term
Description: Actigraphy measurement of average nighttime sleep efficiency (percent time asleep of time in bed): at Week 7 describing the short-term effect of the intervention
Time Frame: Week 7
Population: N=119 participants had at least one time point (week 0, week 7, and/or week 25) with actigraphy data and were included in model to estimate means at week 7 and week 25. Seven had no actigraphy collected: 4 declined to wear the watch; 3 had data that could not be scored due to inconsistent use.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time in bed asleep
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 41 | 41 | 37
percentage of time in bed asleep | 68.03 [62.41 to 73.65] | 70.94 [65.94 to 75.94] | 70.87 [65.94 to 75.8]

24. Secondary Outcome: Objective Measure of Sleep - Long-term
Description: Actigraphy measurement of average nighttime sleep efficiency (percent time asleep of time in bed): at Week 25 describing the long-term effect of the intervention
Time Frame: Week 25
Population: N=119 participants had at least one time point (week 0, week 7, or week 25) with actigraphy data and were included in model to estimate means at week 7 and week 25. Seven had no actigraphy collected: 4 declined to wear the watch; 3 had data that could not be scored due to inconsistent use.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of time in bed asleep
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
Number analyzed (Participants) | 41 | 41 | 37
percentage of time in bed asleep | 68.99 [64.57 to 73.41] | 71.6 [66.77 to 76.43] | 71.57 [65.49 to 77.65]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CBT-I | Medication- Trazodone | Medication- Placebo
All-Cause Mortality (participants affected / at risk) | 2/43 | 3/42 | 3/41
Serious Adverse Events (participants affected / at risk) | 10/43 | 16/42 | 15/41
Other Adverse Events (participants affected / at risk) | 14/43 | 20/42 | 14/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-I (N=43) | Medication- Trazodone (N=42) | Medication- Placebo (N=41)
Hospitalization / Death (Cardiac disorders) | 1 (1) | 8 (13) | 4 (4)
Hospitalization / Death (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalization / Death (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization / Death (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (4)
Hospitalization / Death (Infections and infestations) | 4 (5) | 5 (7) | 7 (9)
Hospitalization / Death (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Hospitalization / Death (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Hospitalization / Death (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization / Death (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization / Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2)
Hospitalization / Death (Surgical and medical procedures) | 3 (3) | 3 (6) | 3 (4)
Hospitalization / Death (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-I (N=43) | Medication- Trazodone (N=42) | Medication- Placebo (N=41)
Hospitalization / Death (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalization / Death (Cardiac disorders) | 2 (3) | 2 (2) | 4 (5)
Hospitalization / Death (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Hospitalization / Death (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization / Death (Gastrointestinal disorders) | 5 (6) | 3 (3) | 3 (3)
Hospitalization / Death (Infections and infestations) | 2 (2) | 3 (3) | 2 (3)
Hospitalization / Death (Injury, poisoning and procedural complications) | 6 (7) | 3 (3) | 4 (7)
Hospitalization / Death (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hospitalization / Death (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4) | 2 (2)
Hospitalization / Death (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1)
Hospitalization / Death (Psychiatric disorders) | 1 (1) | 4 (4) | 0 (0)
Hospitalization / Death (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization / Death (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Hospitalization / Death (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Hospitalization / Death (Surgical and medical procedures) | 0 (0) | 2 (2) | 3 (3)
Hospitalization / Death (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT03534284/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT03534284/ICF_001.pdf